CLINICAL TRIAL: NCT01386060
Title: Mindfulness Meditation in Chronic Stress: Measures of Adherence, Ability & Stress
Brief Title: Mindfulness Meditation in Chronic Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Barry S. Oken, MD, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB7364
Record Dates: First submitted 2011-06-27; First posted 2011-06-30 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Aging
Keywords: Stress; Mindfulness; Meditation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness Meditation Training (Experimental): Participants receive the 6-week meditation training intervention between the 1st and 2nd study visits.
  Interventions: Other: Mindfulness Meditation Training
- Waitlist Control (No Intervention): Participants receive no intervention between the 1st and 2nd study visits. They receive the training between the 2nd and 3rd study visits only.

INTERVENTIONS:
Other: Mindfulness Meditation Training — One-on-one mindfulness meditation training, 6 weeks, 1 1/2 hour training once per week, 30-45 min at-home practice per day.
  Arms: Mindfulness Meditation Training

SUMMARY:
The study purpose is to evaluate efficacy of a mindfulness training intervention and learn about cognitive and physiological markers of stress.

DETAILED DESCRIPTION:
Subjects will first undergo a phone screening, and if eligible, they will complete three study visits at Week 1, Week 8, and Week 15. The study visits involve at-home surveys, voice recordings, physical measures (height, weight, waist-to-hip ratio, and blood pressure), EEG recordings (including recordings of electrodermal activity and heart rate variability), computer tasks, in-lab saliva collection, overnight urine collection, 2-day saliva collection at bed waking, 30 minutes post-waking, afternoon, and bedtime, and a small handheld device that randomly administers eight short assessments in the subjects' natural environment. Subjects will be randomized to receive a 6-week mindfulness meditation course either between the first and second study visits or between the second and third study visits. Participants who receive training during the first and second visits will continue meditating until the third visit. The one-on-one instruction occurs once a week for 1 ½ hours, and participants are asked to listen to guided meditations and do other mindfulness-based tasks on a daily basis between sessions.

ELIGIBILITY:
Inclusion Criteria:

* Ages 50-85
* Good General Health
* Experiencing Stress
* No current meditation practice
* English speaking

Exclusion Criteria:

* Cognitive Impairment
* Neurological Disease
* Major Untreated Depression

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2011-06; Primary Completion 2015-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Changes in Physiological Markers of Stress | Baseline (Week 1) and Visit 2 (Week 8)
  Measure changes in blood pressure, heart rate, heart rate variability, neurological reaction time to visual stimuli, urine, saliva, waist-to-hip ratio, weight, and electrodermal response.

SECONDARY OUTCOMES:
Cognitive Changes | Baseline (Week 1) and Visit 2 (Week 8)
  In-lab cognitive tests measure attention and memory.
Changes in self-reported measures of stress | Baseline (Week 1) and Visit 2 (Week 8)
  A series of questionnaires measure different facets of perceived quality of life and stress

CONTACTS AND LOCATIONS:
Overall Officials: Barry Oken, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- See also: Oregon Center for Complementary and Alternative Medicine — http://www.ohsu.edu/orccamind